CLINICAL TRIAL: NCT05443607
Title: A Prospective Cohort Study Evaluating the Transplacental Transmission of Respiratory Syncytial Virus (RSV) in Pregnant Women and Their Offspring
Brief Title: Transplacental Transmission of RSV (TTRSV)
Status: Active, not recruiting | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-1517
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: SARS CoV 2 Infection; Respiratory Syncytial Virus (RSV); Bronchiolitis; Asthma
Keywords: Fetal blood; COVID-19
MeSH Terms: conditions — COVID-19; Bronchiolitis; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators are extracting RNA for PCR amplification from blood cells, placenta and nasopharyngeal aspirate.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mother infected/newborn not infected
- Mother infected/newborn infected
- Mother not infected/newborn not infected
- Mother not infected/newborn infected

SUMMARY:
Aim 1: To study transplacental transmission of Respiratory Syncytial Virus (RSV) and how this is moderated by other maternal infections during pregnancy

Aim 2: To test maternal blood for presence of RSV-specific immunoglobulins and how this is moderated by other maternal infections during pregnancy

Aim 3: To test cord blood (fetal blood) for presence of RSV-specific immunoglobulins and other common viral pathogens

Aim 4: To perform further tests (Clustered Regularly Interspaced Short Palindromic Repeats (CRISPR), Droplet Digital Polymerase Chain Reaction (ddPCR) and immunoprobing) to confirm the presence of RSV and other common viral pathogens

Aim 5: To follow these newborn infants up to 4 years of age to look for redisposition to respiratory diseases and growth parameters

DETAILED DESCRIPTION:
Patients will be consented at one of two time points during their pregnancy. Option 1: If mothers present or call Obstetrics and Gynecology (OB) with signs or symptoms of an Upper Respiratory Infection (URI) and or a positive SARS-CoV-2 test, the mother's OB will ask if the mother would be interested in hearing about this study at her next prenatal visit if study personnel are not available to discuss the study at the present appointment. If study personnel is available and on-site, they will approach and consent patients who meet criteria after preliminary screening.

Option 2: Mothers who present to labor and delivery and report a history of an URI in the last three weeks and or a history of positive SARS-CoV-2 will be asked by the labor and delivery team or study personnel, if available, about her interest in the study and approached for consent upon admission to labor and delivery. At the time of consent a research blood sample will be drawn if the patient is not already having labs drawn, if the mother agrees.

The additional data collection will be performed electronically. Research staff will contact participants (in person, via email, and via phone, depending on survey timing). REDCap will be used for data collection, with (offline, when necessary) electronic data capture. Participants can access an online version of surveys using their own device or phone, or use tablets provided for the participants for data collection at the hospitals. Participant will have the option to have research staff conduct the question/interview in-person or over the telephone, if this is preferred.

If the mother is enrolled prior to labor, study personnel will then track the enrolled subject's admission to the labor and delivery unit using the electronic health records and regular contact with the OB/GYN service. Study personnel will determine if the subject still meets enrollment criteria after admission to labor and delivery (e.g., baby was carried to at least near full term (34 weeks and beyond) and delivered at either Lakeside Hospital and Clinic or Ochsner Baptist Medical Center). If the patient is still eligible for the study, the study personnel will liaise with bedside nursing to have the maternal research samples collected at the same time standard of care samples are being drawn.

Cord (i.e., fetal) blood, placental tissue, and the newborn naso-pharyngeal aspirate fluid will be collected as early as possible after delivery. All samples will undergo microbiological analyses using Enzyme-Linked Immunoassay (ELISA), Polymerase Chain Reaction (PCR) and CRISPR testing to identify evidence of previous or current infection.

Patients will be given the option of allowing the study team to deidentify and store any remaining maternal and/or infant specimens for additional testing.

Patients will be given the option to allow the study team member to store de-identified remaining maternal and/or infant specimens for future studies.

Patients will be given the option to allow the research team to contact them about their enrollment in any future studies.

All study visits after the collection of biological samples at delivery will be done remotely, through a review of the infant's electronic medical records and questionnaires completed over the phone or via other electronic media (e.g. Zoom) as determined by maternal preference. Mothers will provide information via the use of structured questionnaires delivered and returned by mail every 6 months or by phone based on maternal preference. Telephone interviews and mailed questionnaires will have questions regarding respiratory-related symptoms and diagnoses, allergies, and medications for the index child.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Reported 2 or more signs and symptoms of respiratory infection during pregnancy, including but not limited to: fever, nasal congestion/discharge, cough, and sore throat and/or a positive SARS-CoV-2 test
3. Deliveries at full term or near term (minimum 34 weeks gestation) in Labor and Delivery (L&D) facilities at Tulane Lakeside Hospital and Clinic or Ochsner Baptist Medical Center who were pregnant during RSV season.
4. History negative for Human Immunodeficiency Virus (HIV)
5. No use of immunosuppressive medications/therapies.
6. Singleton gestation;
7. Willing to allow for follow up of the child via their medical record from the time of delivery to 4 years of age.
8. Clearly understands the study procedures and visit schedule, alternative treatments, and risks involved with the study, and voluntarily agrees to participate by giving written informed consent.
9. English or Spanish proficiency

Exclusion Criteria:

1. Under 18 years of age at the time of consent.
2. Gestational age less than 12.0 weeks at the time of consent.
3. Does not report at least 2 of the following signs and symptoms of respiratory infection during pregnancy, including but not limited to: fever, nasal congestion/discharge, cough, and sore throat.
4. Positive medical history for HIV.
5. Current use of immunosuppressive therapies/drugs.
6. Newborn has been diagnosed with congenital abnormality or chronic disease at birth.
7. Unwilling or unable to provide written informed consent.
8. Mother was not pregnant during the RSV season or no positive SARS-CoV-2 test during pregnancy.
9. Subject is unwilling to allow for follow up of the child via medical records from the time of delivery to 4 years of age;
10. Multiple birth;
11. Lacks English or Spanish proficiency

Infants will be excluded from the study in the event of a Serious Adverse Event such as fetal or acute neonatal death (in the delivery room) if the mother does not provide clinical consent for an autopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who plan to deliver at Tulane Lakeside Hospital and Clinic and Ochsner Baptist Medical Center will be considered for inclusion in the study. Pregnant women and their infants who fulfill all inclusion criteria are eligible for participation.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Postnatal respiratory morbidity | 5 Years
  The investigators will monitor the offspring via electronic medical records and mailed questioners to record respiratory symptoms such as upper respiratory infections, cough, wheezing.
Passage of antiviral antibodies from mother to newborn | 5 Years
  The investigators will assess the antiviral protection provided by maternal fetal transport of neutralizing antibodies following maternal vaccination versus natural infection.
Vertical transmission of RSV and/or SARS-COV2 from infected mother to the offspring | 5 Years
  The investigators will use PCR to detect the presence of each virus in maternal blood and cord blood.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Piedimonte, MD, FAAP, FCCP, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - Tulane University Lakeside Hospital, Metairie, Louisiana
  - Ochsner Baptist Hospital, New Orleans, Louisiana